CLINICAL TRIAL: NCT00839189
Title: Safety Study To Determine the Effect of a 10,000 EU Dose of Clinical Center Reference Endotoxin in Allergic and Mildly Asthmatic Adults
Brief Title: Effect of a 10,000 EU Dose of Endotoxin in Allergic and Mildly Asthmatic Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: David Peden, MD/Principal Investigator, UNC Center for Environmental Medicine, Asthma and Lung Biology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 02-1518 (GCRC 1983); NIH HL080337
Record Dates: First submitted 2009-02-06; First posted 2009-02-09 (Estimated); Last update posted 2009-12-09 (Estimated); Status verified 2009-12

CONDITIONS: Rhinitis, Allergic, Perennial; Rhinitis, Allergic, Seasonal; Asthma
Keywords: CCRE; endotoxin; LPS; asthma; allergies; allergic rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Perennial; Rhinitis, Allergic, Seasonal; Asthma; Hypersensitivity; Rhinitis, Allergic | interventions — Endotoxins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Clinical Center Reference Endotoxin (CCRE) — Inhalation of 10,000 EU CCRE
  Other Names: LPS; endotoxin

SUMMARY:
The purposes of this pilot safety study are to identify a dose of inhaled Clinical Center Reference Endotoxin (CCRE) that is well tolerated by allergic subjects that induces measurable increases in neutrophil content of induced sputum that can be employed to screen large populations for susceptibility to the inflammatory effect of inhaled endotoxin.

DETAILED DESCRIPTION:
Twenty-four or forty-eight hours (study day 1) prior to the inhalation challenge, subjects will undergo a physical examination of the ears, nose, throat and chest and will have an assessment of vital signs (temperature, pulse, respiratory rate, blood pressure), oxygen saturation, symptom score assessment and undergo spirometry to rule out acute illness prior to challenge. All female volunteers will undergo a urine pregnancy test. A similar examination will take place immediately prior to inhalation challenge with 10,000 EU of CCRE, as well as 30, 60, 120, 180, 240, 300 and 360 minutes and 24 hours after challenge (with the exception of a pregnancy test which will only be administered prior to sputum induction on study day 1). Induced sputum will be 24 to 48 hours prior to challenge, and again six hours after challenge on Study day 2. Sputum will be analyzed for PMN content, CD14 expression on airway macrophages and monocytes, soluble CD14 levels, cytokine levels in sputum and products of inflammatory cells (eosinophil, cationic protein, myeloperoxidase). Blood will be collected for a CBC and differential when the pre- challenge induced sputum is obtained and again 6 hours after challenge. Subjects will then be escorted to the GCRC for overnight admission. While on the GCRC, vital signs will be obtained every 2 hours till bedtime, then once a shift. Spirometry will not be obtained while the subject is in the GCRC, however the subject will be given symptom scoring cards. The next morning (study day 3) subjects will be discharged and escorted to the CEMALB for a final set of vital signs, spirometry, symptom scoring, and an examination by a study physician.

Each volunteer will be given a symptom scoring sheet for each day up to 96 hours (4 days) after challenge.

Each sheet will include the name and phone number of the study coordinator and study MD. Sample home symptom scoring sheets and instructions are included with this protocol.

Between 48 and 96 hours after challenge, each volunteer will be called to determine their status, inquiring about symptoms, symptom scoring, and need for medication and/or physician visits.

Between 7 and 10 days of the challenge dose, each subject will be asked to return for a study discontinuation visit. At that time temperature, pulse, systolic and diastolic BP, respiratory rate, FVC and FEV1 and SpO2 (oxygen saturation), and symptoms scores will be assessed and, if abnormal, medical evaluation as directed by the study physician will be undertaken.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria
* Specific allergy to at least one of the following allergen preparations: (House Dust Mite f, House dust mite p, Cockroach, Tree mix, Grass Mix, Weed Mix, Mold Mix 1, Mold Mix 2, Rat, Mouse, Guinea Pig, Rabbit, Cat or Dog) confirmed by positive immediate skin test response.
* FEV1 of at least 80% of predicted and FEV1/FVC ratio of at least .75 (without use of bronchodilating medications for 12 hours), consistent with lung function of persons with no more than mild episodic or mild persistent asthma.
* History of nasal allergy, including episodic, perennial, or seasonal sneezing, nasal congestion or cough, or such symptoms associated with specific exposures (such as cat or dog)

Criteria for classification as having asthma with allergic rhinitis vs. allergic rhinitis alone:

* History of episodic wheezing, chest tightness, or shortness of breath consistent with asthma, or physician diagnosed asthma.
* Provocative concentration of methacholine producing a 20% fall in FEV1 (PC20 methacholine) of less than 10 mg/ml by the method used (see below).

Exclusion Criteria:

* Any chronic medical condition considered by the PI as a contraindication to the exposure study including significant cardiovascular disease, diabetes requiring medication, chronic renal disease, or chronic thyroid disease.
* Physician directed emergency treatment for an asthma exacerbation within the preceding 12 months.
* Use of systemic steroid therapy within the preceding 12 months for an asthma exacerbation. All use of systemic steroids in the last year will be reviewed by a study physician.
* Use of inhaled steroids, cromolyn or leukotriene inhibitors (Montelukast or zafirkulast) initiated within the past month (except for use of cromolyn exclusively prior to exercise). Patients must be on a stable regimen of therapy and shown to be stable.
* Use of daily theophylline within the past month.
* Pregnancy or nursing a baby.
* Cigarette smoking > 1 pack per month.
* Nighttime symptoms of cough or wheeze greater than 1x/week at baseline (not during a clearly recognized viral induced asthma exacerbation) which would be characteristic of a person of moderate or severe persistent asthma as outlined in the current NHLBI guidelines for diagnosis and management of asthma.
* Exacerbation of asthma more than 2x/week which would be characteristic of a person of moderate or severe persistent asthma as outlined in the current NHLBI guidelines for diagnosis and management of asthma.
* Daily requirement for albuterol due to asthma symptoms (cough, wheeze, chest tightness) which would be characteristic of a person of moderate or severe persistent asthma as outlined in the current NHLBI guidelines for diagnosis and management of asthma. (Not to include prophylactic use of albuterol prior to exercise).
* Dosing level of an inhaled steroid must be consistent with mild episodic asthma as outlined by the NHLBI NAEPP guidelines. Any dose of inhaled steroid typically used for moderate or severe asthma will result in exclusion from the protocol.
* Viral upper respiratory tract infection within 2 weeks of challenge.
* Any acute infection requiring antibiotics within 2 weeks of challenge.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2002-10; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Magnitude of change in neutrophil content of induced sputum after inhalation of 10,000 EU CCRE | 0-24 hours post challenge

SECONDARY OUTCOMES:
change in PFT's, vital signs and symptom score after inhalation of 10,000 EU of CCRE | 0-24 hours post challenge

CONTACTS AND LOCATIONS:
Overall Officials: David Peden, MD, Principal Investigator — University of North Carolina at Chapel Hill, Dept of Pediatrics / Center for Environmental Medicine, Asthma and Lung Biology
Locations (1):
- UNC Center for Environmental Medicine, Asthma and Lung Biology, Chapel Hill, North Carolina, United States